CLINICAL TRIAL: NCT02590757
Title: Comparison of Non-invasive Ventilation Neurally Adjusted Ventilatory Assist vs. Nasal Continuous Positive Airway Pressure After Extubation in Infants' < 30 Weeks of Gestation: Randomized Controlled Study
Brief Title: Comparison of NIV-NAVA vs. N-CPAP After Extubation in Preterm Infants Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Professor, Director of Neonatal Intensive Care Unit, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1917
Record Dates: First submitted 2015-10-25; First posted 2015-10-29 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Endotracheal Extubation; Infant, Premature
Keywords: non-invasive ventilation; non-invasive neurally adjusted ventilatory assist; nasal continuous positive airway pressure
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIV-NAVA (Active Comparator): Noninvasive ventilation in this group is practiced with NIV-NAVA
  Interventions: Device: NIV-NAVA
- N-CPAP (Active Comparator): Patients in this group will receive nasal continuous positive airway pressure as routinely in neonatal intensive care unit.
  Interventions: Device: N-CPAP

INTERVENTIONS:
Device: NIV-NAVA — Non-invasive neurally adjusted ventilatory assist
  Arms: NIV-NAVA
Device: N-CPAP — Nasal-continuous positive airway pressure
  Arms: N-CPAP

SUMMARY:
This study is a randomized controlled study to compare if a a non-invasive neurally adjusted ventilatory assist (NIV-NAVA) is better than nasal continuous positive airway pressure (N-CPAP) after extubation in infants' < 30 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* postconceptional age less than 30+0 weeks
* infants who fulfill the the criteria for extubation for 6 hours extubation criteria: Ventilator rate ≤ 25 breaths/min, Peak inspiratory pressure (PIP) ≤ 16cmH2O, Fractional inspired oxygen (FiO2) ≤ 0.3

Exclusion Criteria:

* conditions which will decrease life expectancy
* major anomalies which will decrease life expectancy
* any anomalous conditions which involve upper and lower airway
* neuromuscular disease

Ages: 2 Days to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2021-01-23 (Actual)

PRIMARY OUTCOMES:
Extubation failure | extubation - 72 hours
  Failure criteria
  * pH < 7.2 with pCO2 > 70mmHg confirmed by capillary blood gas analysis in spite of maximum settings
  * Severe apnea event requiring bag and mask resuscitation
  * FiO2 >0.6 to maintain SpO2 ≥ 88% after extubation
  * Frequent desaturations (< 85%) ≥ 3/hr not responding to increased ventilatory settings or an increase in Fio2 to 1.0

SECONDARY OUTCOMES:
FiO2 >0.6 to maintain SpO2 ≥ 88% after extubation | extubation - 72 hours
  Participants will be followed for the extubation failure within 3 days after extubation
Severe apnea event requiring bag and mask resuscitation | extubation - 72 hours
  Participants will be followed for the extubation failure within 3 days after extubation
FiO2 >0.6 to maintain SpO2 ≥ 88% after extubation | extubation - 7 days
  Participants will be followed for the extubation failure within 7 days after extubation
pH < 7.2 with pCO2 > 70mmHg confirmed by capillary blood gas analysis in spite of maximum settings | extubation - 7 days
  Participants will be followed for the extubation failure within 7 days after extubation
Severe apnea event requiring bag and mask resuscitation | extubation - 7 days
  Participants will be followed for the extubation failure within 7 days after extubation
Bronchopulmonary dysplasia | postmenstrual age 36 weeks
  Participants will be followed for the duration of hospital stay
Duration of noninvasive ventilation | postmenstrual age 40 weeks (until discharge)
  Participants will be followed for the duration of hospital stay
Duration of inspired oxygen supply | postmenstrual age 40 weeks (until discharge)
  Participants will be followed for the duration of hospital stay
Duration of hospital stay | postmenstrual age 40 weeks (until discharge)
  Participants will be followed for the duration of hospital stay
Adverse events | extubation - 3days
  Participants will be followed for 3 days after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Han-Suk Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin SH, Shin SH, Kim SH, Song IG, Jung YH, Kim EK, Kim HS. Noninvasive Neurally Adjusted Ventilation in Postextubation Stabilization of Preterm Infants: A Randomized Controlled Study. J Pediatr. 2022 Aug;247:53-59.e1. doi: 10.1016/j.jpeds.2022.04.025. Epub 2022 Apr 20. PMID 35460702